CLINICAL TRIAL: NCT05553223
Title: Can Micro-doses of Physical Activity Offset the Negative Cardiovascular Consequences of Being Sedentary in Patients With COPD?
Brief Title: Micro-doses of Physical Activity for COPD
Acronym: COPD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Responsible Party: Principal Investigator, Neil Eves, Professor, University of British Columbia
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: H18-01575
Record Dates: First submitted 2022-06-30; First posted 2022-09-23 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2025-04

CONDITIONS: Chronic Obstructive Pulmonary Disease; Endothelial Dysfunction; Vascular Stiffness; Hypertension; Cardiovascular Diseases
Keywords: Microdoses of Physical Activity; Flow Mediated Dilation; Reactive Hyperemia
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Hypertension; Cardiovascular Diseases; Hyperemia

STUDY DESIGN:
Intervention Model Description: The study will be performed using a prospective randomized crossover design with subjects acting as their own control.
Who Masked: Outcomes Assessor
Masking Description: The investigator who will analyze the primary outcome data will be blinded to the participant and condition.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Microdoses of Activity (Experimental): 5-min bouts of walking will break up 3 hours of sitting at minutes 30, 90 and 150.
  Interventions: Behavioral: Microdoses of activity
- Control (No Intervention): Prolonged sitting (3 hours)

INTERVENTIONS:
Behavioral: Microdoses of activity — Short bouts of low-intensity exercise (walking) will be used to break up prolonged sitting.
  Arms: Microdoses of Activity

SUMMARY:
Chronic obstructive pulmonary disease (COPD) is a disease of the lungs that makes it hard for people to breath. Those with COPD spend considerably more time sitting and lying and less time performing physical activity than healthy individuals. Those who are the most sedentary have a greater risk of heart and blood vessel disease, which may lead to an early death. This project will investigate the effect of sitting still for 3 hours on blood vessel health in individuals with COPD. It will also investigate whether breaking up the amount of time patients sit with regular short bouts of walking (5 minutes each hour) at a comfortable pace chosen by the patient can have a positive effect on maintaining the health of their blood vessels. It is hypothesized that blood vessel health will be worse after 3 hours of sitting compared to when the sitting is broken up by short bouts of walking.

DETAILED DESCRIPTION:
The Purpose of the Study:

The aim of the proposed study is to examine whether regular microdoses of low intensity physical activity (PA) can reduce the vascular dysfunction and adverse cardiovascular consequences associated with being sedentary in patients with COPD.

Hypothesis to be Tested:

Primary Hypothesis: Endothelial function (measured as superficial femoral flow mediated dilation) will be reduced in patients with COPD after 3-hours of prolonged sitting compared to the same duration of sitting interspersed with micro-doses of PA (5 min/hour of walking).

Secondary Hypothesis: Superficial femoral endothelial shear rate and antegrade blood flow will be reduced and retrograde blood flow and arterial stiffness will be increased following prolonged sitting compared to the same duration of sitting interspersed with micro-doses of PA. Mean 24-hour blood pressure will be lower when micro-doses of PA are used to reduce sedentary time.

Exploratory Hypothesis: There will be an increased release of endothelial microparticles (EMP) following prolonged sitting compared to the same duration of sitting interspersed with micro-doses of PA. Furthermore, femoral artery blood antegrade blood flow and shear rate will progressively decline, while retrograde blood flow will increase over each 30 minutes of sitting, but not when regular micro-doses of PA are performed. Flow mediated dilation will progressively decline and (EMP) release will progressively increase with each hour of sitting but not when regular micro-doses of PA are performed.

Justification: The benefits of performing regular moderate-to-vigorous intensity physical activity are well known and are associated with a lower incidence of cardio-metabolic disorders. Patients with chronic obstructive pulmonary disease generally engage in very little moderate to vigorous PA due to exertional dyspnea and typically spend a large portion of each day sitting, reclining or lying down. This increase in sedentary behaviour has been associated with vascular dysfunction, elevated blood pressure and greater risk of cardiovascular mortality in patients with COPD. As sedentary behaviour results in low global blood flow, it is an attractive postulate that one of the detrimental effects of reduced PA may be related to low vascular shear stress. More specifically, reduced shear stress has been documented to impair vascular endothelial function, promote adverse blood flow patterns (i.e. increased retrograde and reduced antegrade flow), increase vascular tone, elevate blood pressure and increase pro-atherosclerotic mediators (i.e. increased circulating levels of endothelial microparticles [EMPs] that are established markers of a dysfunctional and diseased endothelium). Growing evidence suggests that even lower intensity PA or just breaking up sedentary time may have significant health benefits. More specifically, it is feasible that increased blood flow and enhanced shear stress that occurs by moving may have a variety of cardiovascular benefits. Whether reducing sedentary time with regular short bouts (micro-doses) of low intensity PA can offset the adverse vascular consequences of prolonged sedentary behaviour in patients with COPD has not been studied.

Study Design: The study will be performed using a prospective randomized crossover design with subjects acting as their own control. After obtaining informed consent, the first visit will consist of a pulmonary function test to confirm the severity of airflow obstruction. To document current PA levels of subjects and to ensure consistency in PA between the two experimental trials, subjects will be given an accelerometer to measure their habitual physical activity levels and sedentary time on the 5 days before, and on the day of, each experimental trial. Visits 2 and 3 will then be randomized to either: 1) control - sedentary behaviour (either sitting or reclining) for 3 hours or 2) micro-doses - sedentary behavior for 3 hours with 5 minutes of walking every hour. Each visit will be separated by at least 6 days. For 24-hours before, diet will be standardized and patients will be asked to refrain from moderate-to-vigorous PA, alcohol and caffeine. Patients will come fasted (>8hr) for each visit and blood samples and vascular measurements will be made at baseline, and at 1, 2 and 3 hours of prolonged sitting. To further assess blood vessel health 24 hour ambulatory blood pressure measurements will be made following the first vascular assessment at 9am. Statistical Analysis : Data will be assessed for normalcy using a Shapiro-Wilk test. Primary and secondary outcome variables will be analyzed using linear mixed models, with repeated measures of condition (control vs. micro doses) and time (baseline vs post) as fixed factors. If significant interactions are found a Tukey post-hoc analysis will be used. The alpha level for all analysis will be set at 0.05. For the time course data linear mixed models, with repeated measures of condition (control vs. micro doses) and time (0, 1, 2, 3 hours) as fixed factors. Additionally, to assess differences between control and microdoses of PA for mean daytime, night time and nocturnal dipping blood pressures dependent t tests will be used.

ELIGIBILITY:
Inclusion Criteria:

Non-smoking (>6 months) patients with stable moderate-to-severe COPD (post bronchodilator forced expired volume in 1 sec/forced vital capacity<0.7 and <lower limit of normal, 30%<Forced Expired Volume in 1 sec<80% predicted and exacerbation free for >6 weeks) will be recruited for the study.

Exclusion Criteria:

1. performing structured exercise training (or pulmonary rehabilitation)
2. have a history of deep vein thrombosis
3. are on anticoagulant medication
4. have advanced cardiac or cerebrovascular disease (i.e. heart failure, previous stroke or myocardial infarction)
5. have diabetes
6. have musculoskeletal contraindications that limit their ability to perform physical activity
7. vascular ultrasound measurements cannot be obtained.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2022-10-12 (Actual); Primary Completion 2026-09-01 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
Change in superficial femoral artery endothelial function | Within 3 hours of sitting (Day1) or within 3 hours of micro-doses of physical activity (Day 2). Days performed in a randomized order.
  The change in endothelial function (measured by the flow-mediated dilation response to reactive hyperaemia of the superficial femoral artery using ultrasound) from baseline to 3-hours of prolonged sitting in the control condition compared to performing 3-hours of sitting broken up by micro-doses of physical activity.

SECONDARY OUTCOMES:
Difference in 24-hour ambulatory blood pressure between the two conditions | Within 24 hours of sitting (Day 1) or within 24 hours of micro-doses of physical activity (Day 2). Days performed in a randomized order.
  The change in average daytime, night-time and nocturnal-dipping systolic, diastolic and mean blood pressures in the control condition compared to the same pressures after performing 3-hours of sitting broken up by micro-doses of physical activity.
Change in superficial femoral artery blood flow patterns | Within 3 hours of sitting (Day1) or within 3 hours of micro-doses of physical activity (Day 2). Days performed in a randomized order.
  The change in superficial femoral artery shear rate, ante-grade and retrograde flow (measured by femoral ultrasound) from baseline to 3 hours of sitting in the control condition compared to performing 3-hours of sitting broken up by micro-doses of physical activity.

OTHER OUTCOMES:
Time course of change in endothelial function of the superficial femoral artery | Within 1 hour, 2 hours and 3 hours of sitting (Day1) or within 1 hour, 2 hours and 3 hours of micro-doses of physical activity (Day 2). Days performed in a randomized order.
  The time course of change in endothelial function of the superficial femoral artery (as measured by the change in flow mediated dilation at each time point compared to baseline in response to reactive hyperaemia using ultrasound) after each hour of sitting in the control condition compared to the micro-doses of physical activity condition.
Change in central arterial stiffness | Within 3 hours of sitting (Day1) or within 3 hours of micro-doses of physical activity (Day 2). Days performed in a randomized order.
  Change in central arterial stiffness as measured by carotid-femoral pulse wave velocity (using arterial tonometry) from baseline to 3 hours of sitting in the control condition compared to performing 3-hours of sitting broken up by micro-doses of physical activity.
Time course of change in superficial femoral artery blood flow patterns | Within 30, 60, 90, 120, 150 and 180 minutes of sitting (Day1) or within 30, 60, 90, 120, 150 and 180 minutes of sitting broken up by micro-doses of physical activity (Day 2). Days performed in a randomized order.
  The time-course of changes in superficial femoral artery shear rate, antegrade and retrograde flow (measured by ultrasound of the femoral artery) every 30-minutes from baseline to 3 hours of sitting in the control condition compared to compared to every 30-minutes from baseline to 3 hours of sitting broken up by micro-doses of physical activity.
Change in endothelial microparticles | Within 3 hours of sitting (Day1) or within 3 hours of micro-doses of physical activity (Day 2). Days performed in a randomized order.
  The change in endothelial microparticles (CD62E+, CD31+, CD42b-) from baseline to post-3 hours of sitting in the control condition compared to performing 3-hours of sitting broken up by micro-doses of physical activity.

CONTACTS AND LOCATIONS:
Locations (1):
- University of British Columbia, Kelowna, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No
Following study completion, the results will be published with mean data only and participants identities will remain undisclosed.